CLINICAL TRIAL: NCT05051267
Title: Evaluation of the Effectiveness of Mother's Voice, Mothers Embrace and White Noise Methods During Heel Blood Collection
Brief Title: Evaluation of the Effectiveness of Non-pharmacological Methods During Heel Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Uğur Gül, Research Asistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 70904504/43
Record Dates: First submitted 2021-08-31; First posted 2021-09-21 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Infant, Newborn
Keywords: Newborn; Pain; Mother's voice; White noise; Mother Embrace
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Routine Care Group (No Intervention): Before the application, the families will be informed by the researcher and the 'Informed Consent Form' will be signed. After the heel blood procedure, comfort will be provided with gentle touches. For ethical reasons, routine care will be provided when the baby cries.
- Mothers Embrace (Experimental): A mothers embrace is one of the earliest and most common care events that mothers offer to their babies. Close physical contact between mother and baby during hugs can reduce stress by facilitating co-regulation of mother and baby. In a study conducted in Turkey, it was stated that holding the baby on the lap for pain relief in painful interventions is a practical and easy method.
  Interventions: Other: Non-Pharmacological Methods
- White Noise (Experimental): Since white noise is a humming and continuous monotonous sound, it is similar to the sound in the womb (Balci, 2006). It will be explained that this sound is very similar to the sound that the baby hears in the mother's womb by making the white noise recordings listen to the mothers who will have their babies listen to white noise. by Orhan Osman; Dr. From the album 'Kolik', which was created by making use of the album 'The Happiest Baby' prepared by Harvery Karp, which consists only of uterus sounds; The song 'Don't Let Your Baby Cry, PT.2' will be played to babies (Karp, 2015). In addition, infants will be excluded from the study even though they meet the criteria, if they are not sedated, the procedure takes more than 2 minutes, the procedure is disrupted because someone enters the room loudly, or the mother changes the baby's position (Karakoç, & Türker, 2014).
  Interventions: Other: Non-Pharmacological Methods
- Mother's Voice (Experimental): Auditory responses, fetal age 26-28. It develops in the auditory cortex and brain stem in weeks (Eskandari, Keshavarz, & Jahdi, 2010). Hearing is one of the first senses a fetus develops and is 24-33. can recognize and remember the mother's voice after weeks (Djordjevic, 2010 ). The fetus memorizes the musical characteristics of the mother's voice, like tone, by listening to it (Arabin, 2002). It is stated that newborns exposed to their own mother's voice have a lower heart rate, higher sucking rate, a more relaxed appearance, and less crying and body movements (Campbell-Yeo, Fernandes, & Johnston, 2011).
  Interventions: Other: Non-Pharmacological Methods
- Mothers Embrace and White Noise Applied Group (Experimental): One minute after the procedure, the baby's pain score will be evaluated. After the procedure, until the baby returns to basal values, the mother will be asked to hold her baby and the white noise will continue to be listened to. Video and audio recording will continue until the baby's oxygen saturation and heart rate return to pre-procedural basal values. When it returns to basal values, the baby's pain score will be re-evaluated.
  Interventions: Other: Non-Pharmacological Methods
- Mothers Embrace and Mother's Voice Group (Experimental): After the procedure, the baby will continue to listen to the baby who is in the mother's arms. One minute after the procedure, the baby's pain score will be evaluated and the HR and O2 values will be noted. After the procedure, until the baby returns to basal values, the mother will be asked to hold her baby and the mother's voice will continue to be listened to. Video and audio recording will continue until the baby's oxygen saturation and heart rate return to basal values. When it returns to basal values, the baby's pain score will be re-evaluated.
  Interventions: Other: Non-Pharmacological Methods

INTERVENTIONS:
Other: Non-Pharmacological Methods — All of the applications that increase the effectiveness of drugs when used together with analgesics and provide the elimination of pain by releasing our body's natural morphine and endorphins without the use of analgesics are called non-pharmacological treatment.
  Arms: Mother's Voice; Mothers Embrace; Mothers Embrace and Mother's Voice Group; Mothers Embrace and White Noise Applied Group; White Noise

SUMMARY:
Although various pharmacological methods have been used for heel puncture, their effectiveness has not been demonstrated. However, their use is limited due to their sedating effects, toxic effects, and respiratory depressant properties. In this sense, the use of non-pharmacological methods has been examined. Non-pharmacological methods have no side effects, are cheap, and are easily available/applicable. For these reasons, the fact that non-pharmacological methods (appropriate positioning, mother's lap, mother's voice, white noise, oral sucrose, classical music) have been frequently used in recent years, especially during painful interventions. Based on this information, the study was planned as a randomized controlled experimental study to compare the effects of holding the baby in the mother's arms, hearing white noise and mother's voice, or using them in combination during heel blood collection from healthy newborns.

DETAILED DESCRIPTION:
Pain is known to affect individuals of all ages. However, until the 1980s, it was widely believed that newborns were inadequate in perceiving and interpreting pain because their nervous system was not fully developed. Studies conducted after these years have shown that the fetus has all the anatomical structures and functions of the peripheral and central nervous system necessary to perceive and interpret pain from the 20th week. After this information, this issue started to be given more importance in newborns. The most important reason for this is that term and preterm newborns staying in neonatal units experience pain for numerous and very different reasons.

Heel blood sampling, which is widely used for the diagnosis and follow-up of various diseases, causes acute pain in infants. Heel blood collection is more painful than venous blood collection, squeezing is another factor that causes pain. There is not enough data on the chronicity of pain after these procedures. However, the inability to control pain in newborns followed for a long time in health centers increases the risk of chronic pain.

It has been observed that the pain sensitivity of babies who were followed up in the neonatal period and exposed to painful procedures changed in the next period. Therefore, it is very important to measure the infant's perception of pain in order to investigate the causes, mechanisms, and effects of pain. The pain response is very difficult to understand because newborns cannot express themselves verbally. Observation of hormonal, behavioral, and metabolic changes in the body due to pain provides data on the level of response to pain and the effectiveness of treatment. Evaluation of the pain response in the newborn is performed to reveal the pain state, to determine the level of pain, and to understand whether there is a need for intervention. In the routine operation of health centers, it is necessary to give due importance to the evaluation of pain response. It is important to observe the pain conditions as well as the basic vital functions of babies. It has been shown that repetitive heel blood sampling increases sensitivity to pain and decreases the pain threshold. In the light of these findings, it is thought that the heel puncture procedure to collect blood from the heel in the newborn period will have a negative effect on the pain response of the baby in the long term. Although various pharmacological methods have been used for heel puncture, their effectiveness has not been demonstrated. However, their use is limited due to their sedating effects, toxic effects, and respiratory depressant properties. In this sense, the use of non-pharmacological methods has been examined. Non-pharmacological methods have no side effects, are inexpensive, and are easily available/applicable. For these reasons, the fact that non-pharmacological methods (appropriate positioning, mother's lap, mother's voice, white noise, oral sucrose, classical music) have been frequently used in recent years, especially during painful interventions. Based on this information, the study was planned as a randomized controlled experimental study in order to compare the effects of holding the baby in the mother's arms, hearing white noise and mother's voice, or using them in combination during heel blood collection from healthy newborns.

ELIGIBILITY:
Inclusion Criteria:

* Newborns postnatal age is between 1-5 days,
* 37-42. newborns born between gestational weeks,
* Newborns are healthy,
* Babies of mothers without diabetes,
* Newborns were not given any opioid and non-opioid drugs before the application,
* Newborns have been fed at least 30 minutes ago,
* Newborns without any painful interventions other than vitamin K and Hepatitis B injections will be included.
* Mothers can speak and understand Turkish,
* Babies of mothers accepted to participate in the study and written consent form was obtained from them will be included in the study.

Exclusion Criteria:

* Connected to mechanical ventilator,
* Having a neurological disorder,
* Congenital anomaly,
* Having hyperglycemia,
* Having undergone a surgical procedure,
* The baby of a mother is addicted to drugs,
* If the lancet cannot be inserted and removed at once, the baby will be excluded from the study.
* Infants, despite meeting the criteria, will be excluded from the study if the heel blood collection takes more than 2 minutes in total, the procedure is disrupted by someone entering the room loudly, or the mother changes the position of the baby.

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Pain Results | 1 year
  Premature Infant Pain Profile Scale (PIPP)
  PIPP assesses pain with seven indicators. these; three behavioral (forehead wrinkling, squinting eyes, and widening of the nose wings), two physiological (heart rate and oxygen saturation), and two contextual (week of gestation and sleep/wake status) variables (Stevens et al., 1996). Within the scope of the PIPP scale; gestational week, behavioral status, highest heart rate value, lowest oxygen saturation value, forehead wrinkling, squinting eyes, and nose There are 7 items such as expansion on the wings. Each item; is scored as 0, 1, 2, and 3 from best to worst. Premature Infant Pain Profile Scale; Pain is considered mild between 0-6 points, moderate between 7-12 points, and severe between 13-21 points.
Pain Results | 1 year
  Neonatal Infant Pain Scale (NIPS)
  NIPS was developed to assess acute pain. It was developed by Lawrence et al. in 1993. Scoring in NIPS is made according to six categories. These; facial expression, crying, breathing pattern, arms, legs, and alertness. Crying category, three separate points (0-1-2) while others are evaluated with two separate points (0-1). The total score varies between 0-7. The lowest score is "0", while the most severe pain score is "7".
  Lawrence, J., Alcock, D., McGrath, P., Kay, J., MacMurray, S., & Dulberry, C. The development of a tool to assess neonatal pain. 1993; 2(6), 59-66

SECONDARY OUTCOMES:
Physiological Parameters | 1 year
  Oxygen saturation Oxygen values of the newborn before, during and after the procedure
Physiological Parameters | 1 year
  Crying Time The baby's crying time will be noted after receiving heel blood.
Physiological Parameters | 1 year
  Heart Rate Peak Values will be noted by the researcher 1 minute before the procedure, during the heel blood procedure and 1 minute after the procedure.
Physiological Parameters | 1 year
  Basal Values Time

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Gül, Principal Investigator — Akdeniz University Faculty of Nursing
Locations (1):
- Akdeniz University, Kepez, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data sharing plans for the current study are unknown and will be made available at a later date

REFERENCES:
- [Background] Campbell-Yeo M, Fernandes A, Johnston C. Procedural pain management for neonates using nonpharmacological strategies: part 2: mother-driven interventions. Adv Neonatal Care. 2011 Oct;11(5):312-8; quiz pg 319-20. doi: 10.1097/ANC.0b013e318229aa76. PMID 22123399
- [Background] Cignacco E, Hamers JP, Stoffel L, van Lingen RA, Gessler P, McDougall J, Nelle M. The efficacy of non-pharmacological interventions in the management of procedural pain in preterm and term neonates. A systematic literature review. Eur J Pain. 2007 Feb;11(2):139-52. doi: 10.1016/j.ejpain.2006.02.010. Epub 2006 Apr 3. PMID 16580851
- [Background] Apaydin Cirik V, Efe E. The effect of expressed breast milk, swaddling and facilitated tucking methods in reducing the pain caused by orogastric tube insertion in preterm infants: A randomized controlled trial. Int J Nurs Stud. 2020 Apr;104:103532. doi: 10.1016/j.ijnurstu.2020.103532. Epub 2020 Jan 24. PMID 32062050
- [Background] Hermann C, Hohmeister J, Demirakca S, Zohsel K, Flor H. Long-term alteration of pain sensitivity in school-aged children with early pain experiences. Pain. 2006 Dec 5;125(3):278-285. doi: 10.1016/j.pain.2006.08.026. Epub 2006 Oct 2. PMID 17011707
- [Background] Kahraman A, Gumus M, Akar M, Sipahi M, Bal Yilmaz H, Basbakkal Z. The effects of auditory interventions on pain and comfort in premature newborns in the neonatal intensive care unit; a randomised controlled trial. Intensive Crit Care Nurs. 2020 Dec;61:102904. doi: 10.1016/j.iccn.2020.102904. Epub 2020 Jul 9. PMID 32653359
- [Background] Karakoc A, Turker F. Effects of white noise and holding on pain perception in newborns. Pain Manag Nurs. 2014 Dec;15(4):864-70. doi: 10.1016/j.pmn.2014.01.002. Epub 2014 Feb 20. PMID 24559599
- [Background] Kucukoglu S, Aytekin A, Celebioglu A, Celebi A, Caner I, Maden R. Effect of White Noise in Relieving Vaccination Pain in Premature Infants. Pain Manag Nurs. 2016 Dec;17(6):392-400. doi: 10.1016/j.pmn.2016.08.006. Epub 2016 Oct 15. PMID 27751753
- [Background] Leng HY, Zheng XL, Zhang XH, He HY, Tu GF, Fu Q, Shi SN, Yan L. Combined non-pharmacological interventions for newborn pain relief in two degrees of pain procedures: A randomized clinical trial. Eur J Pain. 2016 Jul;20(6):989-97. doi: 10.1002/ejp.824. Epub 2015 Dec 18. PMID 26685099
- [Background] Neu M, Robinson J, Schmiege SJ. Influence of holding practice on preterm infant development. MCN Am J Matern Child Nurs. 2013 May-Jun;38(3):136-43. doi: 10.1097/NMC.0b013e31827ca68c. PMID 23625100
- [Background] Ahmadi M, Toghyani R, Shahidi S, Izadi M, Merasi MR, Agdak P, Meshkaty M, Nikkhahfard M. The study of Prevalence of Antigen HBs Positive and High-risk Behaviors in Pregnant Women Referring to Urban Health Centers of Isfahan Province in 2009. Iran J Nurs Midwifery Res. 2011 Winter;16(1):1-8. PMID 21772915
- [Background] Stevens B, Johnston C, Petryshen P, Taddio A. Premature Infant Pain Profile: development and initial validation. Clin J Pain. 1996 Mar;12(1):13-22. doi: 10.1097/00002508-199603000-00004. PMID 8722730
- [Background] Walter-Nicolet E, Annequin D, Biran V, Mitanchez D, Tourniaire B. Pain management in newborns: from prevention to treatment. Paediatr Drugs. 2010 Dec 1;12(6):353-65. doi: 10.2165/11318900-000000000-00000. PMID 21028915
- [Background] Yin T, Yang L, Lee TY, Li CC, Hua YM, Liaw JJ. Development of atraumatic heel-stick procedures by combined treatment with non-nutritive sucking, oral sucrose, and facilitated tucking: a randomised, controlled trial. Int J Nurs Stud. 2015 Aug;52(8):1288-99. doi: 10.1016/j.ijnurstu.2015.04.012. Epub 2015 Apr 23. PMID 25939641
- [Background] Anand KJ, Coskun V, Thrivikraman KV, Nemeroff CB, Plotsky PM. Long-term behavioral effects of repetitive pain in neonatal rat pups. Physiol Behav. 1999 Jun;66(4):627-37. doi: 10.1016/s0031-9384(98)00338-2. PMID 10386907